CLINICAL TRIAL: NCT03227380
Title: Morphologic Study of the Intersegmental Plane After Fully Thoracoscopic Segmentectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: THO-2016-01
Record Dates: First submitted 2017-06-19; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Video-assisted Thoracoscopic Surgery (VATS); Segmentectomy
MeSH Terms: interventions — Contrast Media

STUDY DESIGN:
Intervention Model Description: patients undergo anatomic segmentectomy by video-assisted thoracoscopic surgery (VATS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiological evaluation (Other): to explore by thoracic densitometry with contrast the spared segments after stapling of the intersegmental plan following a thoracoscopic segmentectomy
  Interventions: Other: thoracic densitometry with contrast

INTERVENTIONS:
Other: thoracic densitometry with contrast — injected CT scan at 3 or 6 months after segmentectomy VATS

SUMMARY:
The objective of this study is to determine whether stapling adversely affects the pulmonary parenchyma and the vascularisation of the adjacent segments. The aim of our work is to explore by thoracic densitometry with contrast the spared segments after stapling of the intersegmental plan following a thoracoscopic segmentectomy, 3 or 6 months post-surgery. the investigator will assess venous drainage and the arterial vascularisation of the remaining segments, possible modifications of the adjacent parenchyma and whether there is a defect of pleuro-pulmonary adhesion (residual pneumothorax).

DETAILED DESCRIPTION:
Scheduled anatomical segmentectomies are increasingly popular, due to the development of minimally invasive techniques, the increased incidence of early-stage tumours, and the possibility of caring for patients with compromised health and/or limited respiratory function without compromising the oncological outcome, compared to current alternatives such as stereotactic ablative radiotherapy (1).

One of the challenges in the development of the thoracoscopic segmentectomy technique we have published (2-5) is the orientation (6-7) and the division of the intersegmental plane, by contrast to segmentectomy by thoracotomy where this is helped by palpation and the manual traction which can be used on the segment, along the intersegmental vein. The most commonly used technique to separate two adjacent segments remains stapling, despite its high cost and sometimes giving a less anatomical section, with a risk to encroach on the intersegmental vein. Moreover, there can be a partial plicator of the spared segment(s) which could in theory make them less functional.

We have however shown that the postoperative morbidity and mortality rates were much lower than that of patients who had a thoracotomy, dropping from 42% for thoracotomies to 16% for thoracoscopies, the surgical approach being an independent predictive factor for postoperative complications (8).

ELIGIBILITY:
Inclusion Criteria:

* Enrolment in the study will be offered to all patients having undergone a programmed scheduled video-assisted thoracoscopic segmentectomy, whatever the aetiology.
* Men or women aged 18 years or greater
* Absence of severe hepatic insufficiency
* signed and dated informed consent
* candidate for segmentectomy
* Registration in a national healthcare system.
* Women of child-bearing age using effective oral or barrier contraception

Exclusion Criteria:

* Proven intolerance to iodinated contrast agents
* Know allergy or non-controlled asthma - pregnancy
* Severe hepatic insufficiency (creatinine clearance < 30ml/min, by Cockroft's method)
* Pregnant or breastfeeding women
* Patients under trusteeship or curators
* Diabetic patients or patients receiving oral antidiabetic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-02-20 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
The measure of the remaining segments after stapling the intersegmental plane by injected CT scan | 3 or 6 months after surgery
  The aim of investigators work is to explore by thoracic densitometry with contrast the spared segments after stapling of the intersegmental plan following a thoracoscopic segmentectomy, from 3 to 6 months post-surgery. The investigators will assess venous drainage and the arterial vascularisation of the remaining segments, possible modifications of the adjacent parenchyma and whether there is a defect of pleuro-pulmonary adhesion (residual pneumothorax).
  The radiological evaluation criteria will be:
  * Presence and quantification of a defect in pulmonary expansion (residual pneumothorax)
  * Abnormal venous and arterial vascularisation of the remaining segments
  * Defect of the pulmonary parenchyma in contact with the staples line (atelectasis, vascularisation defect)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Mutualiste montsouris, Paris
  - Institut mutualiste montsouris, Paris

IPD SHARING:
Plan to Share IPD: Undecided